CLINICAL TRIAL: NCT07307573
Title: A Remotely Supported Pediatric Simulation-Based Procedural Training Curriculum for EMS Clinicians: Partnering PECCs and Pediatric Experts at a Distance
Brief Title: A Remotely Supported Pediatric Simulation-Based Procedural Training Curriculum for EMS Clinicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-0172; 2UL1TR001425-05A1 (NIH)
Record Dates: First submitted 2025-12-23; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Education; Emergency Medical Services
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: all participants received the same educational intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- educational intervention (Experimental): received training and submitted video on each procedure
  Interventions: Behavioral: education

INTERVENTIONS:
Behavioral: education — pediatric emergency care coordinator provided education on each procedure performed

SUMMARY:
The purpose of this study is to study and compare the efficacy and feasibility of a remotely supported simulation-based procedural curriculum for Emergency Medical Services (EMS) clinicians.

DETAILED DESCRIPTION:
This study transitioned a previously reported, traditional, simulation-based training curriculum delivered by on-site pediatric simulation experts, into a program delivered by agency Pediatric Emergency Care Coordinators (PECCs) supported by remote pediatric experts. The PECCs delivered the curriculum on site, and submitted first-person-view videos captured using a head-mounted camera of three procedures (bag-valve mask [BVM] ventilation, supraglottic device [SGD] insertion, and intraosseous [IO] catheterization) to pediatric education experts who provided scoring and feedback to the participants. The team tracked scores for all three procedures during the study period, compared scores to the previous study's, and solicited feedback from the PECCs and participants regarding these educational methods.

ELIGIBILITY:
Inclusion Criteria:

* all full-time or part-time EMS clinicians at the recruited agencies with BVM ventilation, SGD placement, and/or IO catheterization within their scope of practice

Exclusion Criteria:

* no procedures of interest within scope of practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
intraosseous (IO) catheterization procedural outcome score | participants submitted 1-2 procedural videos based on training date during the 1-year study period
  The IO assessment tool was adapted from a previously validated simulation assessment tool. The score ranged from 0-12, with higher score demonstrating better performance. Participants submitted videos for review, which were scored by trained video reviewers using the assessment tool based on a corresponding data dictionary. Scores were then aggregated for analysis.
bag valve mask (BVM) ventilation procedural outcome score | participants submitted 1-2 procedural videos based on training date during the 1-year study period
  The BVM assessment tool was adapted from a previously validated simulation assessment tool. The score ranged from 0-12, with higher score demonstrating better performance. Participants submitted videos for review, which were scored by trained video reviewers using the assessment tool based on a corresponding data dictionary. Scores were then aggregated for analysis.
supraglottic device (SGD) placement procedural outcome score | participants submitted 1-2 procedural videos based on training date during the 1-year study period
  The SGD assessment tool was modified from a prior psychomotor examination checklist used by the National Registry of Emergency Medical Technicians. The score ranged from 0-14, with higher score demonstrating better performance. Participants submitted videos for review, which were scored by trained video reviewers using the assessment tool based on a corresponding data dictionary. Scores were then aggregated for analysis.

SECONDARY OUTCOMES:
qualitative feedback regarding the curriculum | 1 year study period
  Feedback regarding the curriculum and educational experience was solicited via e-mail from participants at time of score reporting. Similar feedback was solicited via e-mail from educators throughout the study period during scheduling or troubleshooting correspondences. Comments were tabulated and summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hoon Lee, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SH, Riney LC, Merkt B, McDonough SD, Baker J, Boyd S, Zhang Y, Geis GL. Improving Pediatric Procedural Skills for EMS Clinicians: A Longitudinal Simulation-Based Curriculum with Novel, Remote, First-Person-View Video-Based Outcome Measurement. Prehosp Emerg Care. 2024;28(2):352-362. doi: 10.1080/10903127.2023.2263555. Epub 2024 Feb 1. PMID 37751212